CLINICAL TRIAL: NCT00781612
Title: An Open-Label, Multicenter Extension Study of Trastuzumab Emtansine Administered as a Single Agent or in Combination With Other Anti-Cancer Therapies in Patients Previously Enrolled in a Genentech and/or F. Hoffmann-La Roche Ltd-Sponsored Trastuzumab Emtansine Study
Brief Title: A Safety Extension Study of Trastuzumab Emtansine in Participants Previously Treated With Trastuzumab Emtansine Alone or in Combination With Other Anti-Cancer Therapy in One of the Parent Studies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDM4529g; BO25430 (Other: Hoffmann-La Roche); 2010-021067-32 (EudraCT Number); 2023-503479-79-00 (Other: EU CT)
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Docetaxel; Paclitaxel; pertuzumab; Trastuzumab; Ado-Trastuzumab Emtansine; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trastuzumab Emtansine (Experimental): Participants will receive trastuzumab emtansine either as a single agent or in combination with other anti-cancer therapy (atezolizumab, paclitaxel, trastuzumab and docetaxel). Participants will receive the same dose and schedule on Cycle 1, Day 1 at which it was given at the end of the parent study. Study drug will be administered in 21-day cycles or weekly, depending on the schedule used in the parent study. Participants will receive study treatment until disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Drug: Paclitaxel; Drug: Pertuzumab; Drug: Trastuzumab; Drug: Trastuzumab Emtansine; Drug: Atezolizumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel will be administered as per local prescribing information.
Drug: Paclitaxel — Paclitaxel will be administered as per local prescribing information.
Drug: Pertuzumab — Pertuzumab will be administered intravenously at a dose of 420 milligrams (mg) no more frequently than every 3 weeks (Q3W) (or as directed in the parent study protocol if less than Q3W).
  Other Names: Perjeta
Drug: Trastuzumab — Trastuzumab will be administered as per local prescribing information.
  Other Names: Herceptin
Drug: Trastuzumab Emtansine — Trastuzumab emtansine will be administered as intravenous (IV) infusion. Participants on weekly dosing schedule of trastuzumab emtansine in parent study, may switch to Q3W schedule as per the clinical judgment of the investigator. The starting dose of Q3W schedule must not exceed 3.6 milligrams per kilograms (mg/kg).
  Other Names: Kadcyla; T-DM1
Drug: Atezolizumab — Atezolizumab will be administered at a dose of 1200 mg by IV infusion every three weeks (Q3W)
  Other Names: Tecentriq

SUMMARY:
This is a global, multicenter, open-label safety extension study. Participants receiving single-agent trastuzumab emtansine or trastuzumab emtansine administered in combination with other anti-cancer therapies in a Genentech / Roche-sponsored parent study who are active and receiving benefit at the closure of parent study are eligible for continued treatment in this study.

ELIGIBILITY:
Inclusion Criteria:

* Completed single-agent trastuzumab emtansine or combination trastuzumab emtansine treatment in the parent study or who continue to receive single-agent trastuzumab emtansine or combination trastuzumab emtansine treatment at the time of the parent study closure and received the last study drug dose within the 6 weeks (42 days) prior to the first dose of study therapy on the extension study or Continue to receive treatment in the control arm of study BO21976/TDM4450g (NCT00679341) at the time of the parent study closure if the participant received the last dose of control arm study drug within the 6 weeks (42 days) prior to the first dose of control arm study therapy in the extension study
* Participants in the control arm from Study BO21976/TDM4450g whose disease progression has occurred during the transition interval between the parent study and this extension study may initiate trastuzumab emtansine treatment at the time of enrollment into study TDM4529g (NCT00781612)
* Expectation by the investigator that the participant may continue to benefit from additional single-agent trastuzumab emtansine or combination trastuzumab emtansine treatment or Expectation of the investigator that the participant may continue to benefit from control arm treatment as given in study BO21976/TDM4450g and at the time of disease progression may benefit from single-agent trastuzumab emtansine treatment
* Women of childbearing potential and men with partners of childbearing potential, must be willing to use a highly effective form of non-hormonal contraception or two effective forms of non-hormonal contraception by the participants and/or partner, and to continue the use of contraception for the duration of study treatment and for at least 5 months after the final dose of atezolizumab (if applicable) or 7 months after the final dose of trastuzumab, trastuzumab emtansine or pertuzumab, whichever is later. Women must refrain from donating eggs during this same period
* Male participants whose partners are pregnant should use condoms for the duration of the pregnancy. Men must refrain from donating sperm during this same period

Exclusion Criteria:

* AEs leading to single-agent trastuzumab emtansine or combination trastuzumab emtansine treatment discontinuation in the parent study
* Ongoing SAEs from the parent study
* Progressive disease on single-agent trastuzumab emtansine or a trastuzumab emtansine-containing regimen during the parent study or before starting the extension study, with the exception of participants from study TDM4688g (NCT00943670) with early disease progression who went on to receive pertuzumab + trastuzumab emtansine treatment and have not experienced further disease progression on the combination regimen
* Peripheral neuropathy of Grade greater than or equal to (>/=) 3 per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 3.0, 4.0 or 5.0, as utilized in the parent study
* History of symptomatic congestive heart failure ([CHF]; New York Heart Association [NYHA] Classes II-IV), ventricular arrhythmia requiring treatment, current unstable angina, or history of myocardial infarction within 6 months prior to study entry
* Severe dyspnea at rest due to complications of advanced malignancy or current requirement for continuous oxygen therapy
* Current severe, uncontrolled systemic disease (for example [e.g.] clinically significant cardiovascular, pulmonary, or metabolic disease)
* Major surgical procedure or significant traumatic injury within 28 days prior to study entry or anticipation of the need for major surgery during the course of study treatment
* Current pregnancy or lactation
* History of receiving any investigational treatment or other systemic therapy directed at controlling cancer (e.g., chemotherapy, trastuzumab, etc.) since the participant's last study drug dose in the parent study
* History of hypersensitivity with previous trastuzumab emtansine or any agent used with trastuzumab emtansine in the parent study, precluding further dosing
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2008-10-16 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to 30 days after last dose of study drug administration (up to approximately 14 years)
Percentage of Participants With Adverse Events Leading to Study Treatment Discontinuation or Dose Reduction | Baseline up to 30 days after last dose of study drug administration (up to approximately 14 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (178):
- United States (49):
  - City of Hope National Medical Center, Duarte, California
  - Can Care Assoc Med Group Inc, Redondo Beach, California
  - Univ of Calif, San Francisco, San Francisco, California
  - Central Coast Medical Oncology, San Luis Obispo, California
  - UCLA Oncology Office, Santa Monica, California
  - Stanford Cancer Institute, Stanford, California
  - Kaiser Permanente - Walnut Creek, Walnut Creek, California
  - Univ of Colorado Canc Ctr, Aurora, Colorado
  - University of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Center - Denver, Denver, Colorado
  - Christina Care Institutional Review Board, Newark, Delaware
  - Florida Cancer Specialists, Fort Myers, Florida
  - Memorial Cancer Institute at Memorial West, Pembroke Pines, Florida
  - Florida Cancer Specialists (St. Petersburg ? St. Anthony?s Professional Building), St. Petersburg, Florida
  - Florida Cancer Specialists - Tampa (Dr. MLK Blvd), Tampa, Florida
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Kootenai Cancer Center, Post Falls, Idaho
  - Loyola University Med Center, Maywood, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Hematology-Oncology, Bettendorf, Iowa
  - Oncology Assoc of Cedar Rapids, Cedar Rapids, Iowa
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Johns Hopkins Univ Med Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology Hematology, Pa, Minneapolis, Minnesota
  - University of Minnesota., Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Mercy Clinic Cancer & Hematology, Springfield, Missouri
  - St. John's Mercy Medical Ctr, St Louis, Missouri
  - Comp Cancer Centers of Nevada, Las Vegas, Nevada
  - St. Barnabas Health Care Sys, Livingston, New Jersey
  - Clinical Research Alliance, Lake Success, New York
  - NS-Long Island Jewish Hlth Sys, Lake Success, New York
  - Laura and ISAAC Perlmutter Cancer Center at NYU Langone., New York, New York
  - Carolina Oncology Specialists, PA - Hickory, Hickory, North Carolina
  - The Mark H. Zangmeister Ctr, Columbus, Ohio
  - Northwest Cancer Specialists - Portland (N Broadway), Portland, Oregon
  - Sarah Cannon Research Institute / Tennessee Oncology, Chattanooga, Tennessee
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology, Bedford, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - USO, Plano, Texas
  - Cancer Therapy & Research Center, San Antonio, Texas
  - USO - Tyler Cancer Ctr, Tyler, Texas
  - Uni of Washington Medical Center, Seattle, Washington
  - Univ of WA Medical Center, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Australia (2):
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Peter MacCallum Cancer Center, Melbourne, Victoria
- Belgium (2):
  - UZ Gent, Ghent
  - ZAS Sint Augustinus Wilrijk, Pharmacy, Wilrijk
- Brazil (6):
  - Clinica de Oncologia de Porto Alegre - CliniOnco, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
  - Instituto Nacional de Cancer - INCa, Rio de Janeiro
- Bulgaria (2):
  - Complex Oncology Center - Plovdiv First Internal Chemotherapy Department, Plovdiv
  - SHATO - Sofia, Sofia
- Canada (4):
  - BC Cancer ? Kelowna (Sindi Ahluwalia Hawkins Centre), Kelowna, British Columbia
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Québec ? Hôpital du Saint-Sacrement / ONCOLOGY, Québec
- Fundacion Arturo Lopez Perez, Santiago, Chile
- China (10):
  - The Affiliated Hospital of Military Medical Sciences(The 307th Hospital of Chinese PLA), Beijing
  - Beijing Cancer Hospital, Beijing
  - the First Hospital of Jilin University, Changchun
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Cancer Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
- Czechia (2):
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Poliklinika Vseobecne Fakultni Niemocnice, Prague
- Denmark (2):
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense
  - Vejle Sygehus, Vejle
- France (8):
  - Centre Francois Baclesse, Caen
  - Centre Georges Francois Leclerc, Dijon
  - Institut Paoli Calmettes, Marseille
  - Institut régional du Cancer Montpellier, Montpellier
  - Hopital Tenon, Paris
  - Institut Curie, Paris
  - Institut Curie - Hopital Rene Huguenin, Saint-Cloud
  - Ico Rene Gauducheau, Saint-Herblain
- Germany (5):
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - Frauenarzt-Zentrum Zehlendorf an der Teltower Eiche, Berlin
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Rotkreuzklinikum München, München
  - Klinikum der Universität München, München
- Grupo Angeles, Guatemala City, Guatemala
- Queen Mary Hospital, Hong Kong, Hong Kong
- Hungary (3):
  - Szent Margit Hospital, Budapest
  - Debreceni Egyetem, Klinikai Kozpont, Onkologiai Klinika, Debrecen
  - Markusovszky Hospital, Szombathely
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Ctr, Tel Aviv
- Italy (12):
  - Ospedale San Carlo, Potenza, Basilicate
  - Campus Universitario S.Venuta, Catanzaro, Calabria
  - Istituto Nazionale Tumori Irccs Fondazione g. PASCALE, Napoli, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - Ospedale Regionale Di Parma, Parma, Emilia-Romagna
  - RCCS - Centro di Riferimento, Aviano (PN), Friuli Venezia Giulia
  - Azienda Ospedaliero-Universitaria Dipartimento Interaziendale Di Oncologia, Udine, Friuli Venezia Giulia
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo, Candiolo, Piedmont
  - Ospedale Civile, Sassari, Sardinia
  - Humanitas Istituto Clinico Catanese S.p.A, Misterbianco (CT), Sicily
- Japan (2):
  - Hiroshima University Hospital, Hiroshima
  - Hyogo Cancer Center, Hyōgo
- Mexico (3):
  - Centro de Investigacion, Acapulco de Juárez, Guerrero
  - Instituto Nacional de Cancer, D.F., Mexico CITY (federal District)
  - Consultorio de Medicina Especializada, Distrito Federal
- Auckland city hospital, Auckland, New Zealand
- Private Health Organization Acibadem Sistina Hospital, Skopje, North Macedonia
- Oslo Universitetssykehus HF, Oslo, Norway
- The Panama Clinic, Panama City, Panama
- Peru (2):
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Instituto, Lima
- Philippines (3):
  - Cebu Cancer Institute, Cebu City
  - Veterans Memorial Medical Ctr, Quezon City
  - Cardinal Santos Medical Center, San Juan City
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - ?wi?tokrzyskie Centrum Onkologii, Kielce
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Klinika Onkologii, Otwock
  - Wielkopolskie Centrum Onkologii, Poznan
  - Wojewódzki Szpital Specjalistyczny Nr 3, Rybnik
  - Narodowy Instytut Onkologii im. M.Sklodowskiej-Curie, Warsaw
- Portugal (3):
  - Hospital da Luz, Lisbon
  - Centro Hospitalar do Porto ? Hospital de Santo António, Porto
  - IPO do Porto, Porto
- Russia (7):
  - Bashkirian Republican Clinical Oncology Dispensary, Ufa, Bashkortostan Republic
  - SBIH Republican Clinical Oncological Dispensary of the MoH of Republic Bashkortostan, Ufa, Bashkortostan Republic
  - City Clinical Oncology Hospital, Moscow, Moscow Oblast
  - Blokhin Cancer Research Center, Moskva, Moscow Oblast
  - FSBI?National Medical Research Center of Oncology named after N.N.Petrov? MHRF, Saint Petersburg, Sankt-Peterburg
  - City Oncology Dispensary, Saint Petersburg, Sankt-Peterburg
  - SBI of Healthcare of Stavropol region Stavropol Regional Clinical Oncology Dispensary, Stavropol
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Korea (7):
  - Kyungpook National University Medical Center, Daegu
  - National Cancer Center, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (11):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital de Jerez de la Frontera, Jerez de la Frontera, Cadiz
  - Hospital de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital del Mar, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Hospital San Pedro De Alcantara, Cáceres
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- Universitätsspital Zürich, Zurich, Switzerland
- Taiwan (2):
  - Chi-Mei Medical Center, Tainan
  - National Taiwan Uni Hospital, Taipei
- Thailand (2):
  - Bumrungrad International Hosp, Bangkok
  - Rajavithi Hospital, Bangkok
- United Kingdom (12):
  - Ninewells Hospital, Dundee
  - Western General Hospital, Edinburgh
  - Diana Princess of Wales Hosp., Grimsby
  - Royal Lancaster Infirmary, Morecambe Bay Hospitals Nhs Trust, Lancaster
  - Royal Free Hospital, London
  - Christie Hospital NHS Trust, Manchester
  - Mount Vernon Hospital, Middlesex
  - Nottingham City Hospital, Nottingham
  - Poole General Hospital, Poole
  - Queen's Hospital, Romford
  - Abertawe and Bro Morgannwg NHS Trust, Swansea
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing